CLINICAL TRIAL: NCT03443271
Title: Effect of Transversus Abdominis Plane (TAP) Block and the Perioperative Stress Response: Randomized Control Trial in Patient Undergoing Total Abdominal Hysterectomy in a Tertiary Care Hospital of Pakistan
Brief Title: Effect of TAP Block on Stress Hormones
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Samina Ismail, Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4718-Ane-ERC-17
Record Dates: First submitted 2018-01-26; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Abdominal Hysterectomy; Postoperative Pain
Keywords: transversus abdominis plane block; abdominal hysterectomy; stress response
MeSH Terms: conditions — Pain, Postoperative; Fractures, Stress

STUDY DESIGN:
Intervention Model Description: Prospective double blind randomized control trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be randomly allocated in equal groups of 25 each to undergo TAP block (T group) with 20ml of 0.25% bupivacaine per side or TAP block with 20 ml of normal saline on both sides, which will be the control group (C group). The allocation sequence will be generated by a random number table, and group allocation will be concealed in sealed, opaque envelopes, which will not be opened until patient consent will be obtained. The process of randomization and blinding will be done by the clinical trial unit and according to the group allocation; pre-formed sterile syringes will be dispensed by the clinical trial unit to anesthesiologist performing the TAP block. The anesthesiologist performing the TAP block, patients and staff providing postoperative care will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T (TAP Block with Bupivicaine) (Experimental): Ultrasound guided TAP block will be performed in this group. Bupivicaine 0.25 % 20 ml will be administered in the block on either side.
  Interventions: Procedure: TAP Block with Bupivicaine
- Group C (TAP Block with Placebo drug) (Placebo Comparator): Ultrasound guided TAP block will be performed in this group. 0.9 % Saline 20 ml will be administered in the block on either side.
  Interventions: Procedure: TAP Block with Placebo drug

INTERVENTIONS:
Procedure: TAP Block with Bupivicaine — Ultrasound guided TAP block will be performed and patient will be administered 20 ml of 0.25 % Bupivicaine on each side.
  Arms: Group T (TAP Block with Bupivicaine)
Procedure: TAP Block with Placebo drug — Ultrasound guided TAP block will be performed and patient will be administered 20 ml of 0.9% Saline on each side.
  Arms: Group C (TAP Block with Placebo drug)

SUMMARY:
Random allocation of patients in two groups; Tap block group (T group) and control group (C group). All patients will receive standard general anesthesia and postoperative pain management. The TAP group patient will receive ultrasound guided (US) TAP block with 20 cc of 0.25% of bupivacaine and control group will receive 20cc of normal saline. TAP block in both groups will be performed with US guidance and the study drug will be injected after complete visualization of the needle tip between the internal oblique and the transversus abdominis muscles.

Venous blood samples (5 ml for each time) for metabolic and stress hormones, including, Serum cortisol and nor-epinephrine will be collected before anesthesia at the time of cannulation (T1),60 minutes after incision(T2), 6hrs (T3)and 12 h (T4) after the surgery.

Postoperatively patient will be put on patient controlled intravenous infusion of nalbuphine

DETAILED DESCRIPTION:
Total abdominal hysterectomy (TAH) is a commonly performed major surgical procedure that results in substantial postoperative pain and discomfort. It has been shown that surgical pain and trauma can lead to a number of hormonal changes initiated by the neuronal activation of the hypothalamic pituitary-adrenal axis and the sympathetic nervous system, which can have a detrimental effect on the patient. Strenuous effort has been made to inhibit the stress response to surgery and evaluate its outcome.

It has been shown that this stress response is influenced by the mode of anesthesia and postoperative analgesia. A surgery induced stress response blunted by regional technique and the potential benefits of regional analgesia on surgical outcome are still under scrutiny. Among the postoperative analgesic technique, epidural analgesia has shown to significantly abolish the perioperative stress responses after number of surgeries including hysterectomy. In Pakistan only a small proportion of women wants to avail the epidural service due to fears and misconception.

Another modality of regional technique that has gained popularity as a part of multimodal analgesia is transversus abdominis plane (TAP) block. It is a newly developed block involving the nerves of the anterior abdominal wall. The abdominal wall sensory afferents course through the transversus abdominis plane superficial to the transversus abdominis muscle. An important component of the pain experienced by patients after abdominal surgery derives from the abdominal wall incision.

The efficacy of the TAP block in providing postoperative analgesia as a part of multimodal analgesia has been demonstrated in number of surgeries including colonic resection surgery, caesarean delivery, radical prostatectomy and also hysterectomy. In literature search investigators did not find any clinical study that has been carried out to see the effect of TAP block on stress response after hysterectomy. This study is designed to test the hypothesis that the TAP block, as part of a multimodal analgesic regimen, would attenuate stress response after TAH when compared with placebo. The investigators will also see any difference in postoperative pain and rescue analgesic demands and side effects among patients.

Rationale for the study

Background information:

Failure to adequately control postoperative acute pain can have a number of unwanted physiological and psychosocial consequences for the patient including dissatisfaction, myocardial problems, prolonged hospital stay and even the potential progression to chronic pain. Pain associated with abdominal surgery can be very severe and can lead to a number of hormonal changes initiated by the neuronal activation of the hypothalamic pituitary-adrenal axis and the sympathetic nervous system, which can have a detrimental effect on the patient.

Current postoperative analgesic regimens rely heavily on systemic opioid analgesics which are associated with a number of undesirable side effects including nausea, vomiting, constipation, respiratory depression, and many others. In addition developing countries like Pakistan have limited supply of good quality opioids ,thus safer alternatives need to be evaluated. As a result postoperative pain management in a developing country like Pakistan has been less than suboptimal and barriers include general lack of resources in terms of personnel, drug availability and basic equipment

It has been observed that in developing countries only 45% of anesthetist had ready access to morphine and pethidine. Currently, the cost of importing morphine to developing countries is disproportionately high. A survey of opioid costs in 2003 showed that opioid drugs were up to 10 times more expensive in the developing world than in the developed world, after adjustment for differences in gross domestic product. Therefore in order to find the alternatives; local anaesthetic techniques by means of regional analgesic technique can provide excellent postoperative pain relief and their use should be encouraged whenever possible. There is a need to find techniques to improve postoperative analgesia which will decrease the requirement for opioids, are safe, cost effective, easy to perform and acceptable to patients.

TAP block a form of regional analgesia has been investigated as a part of multimodal analgesia and has shown promising result in decreasing the pain scores and opioid consumption but its role in inhibiting the surgical stress response is still not known. TAP block has been practiced at Aga Khan University hospital (AKUH) since 2012 now, but no data regarding its effect on stress hormones has been collected.

Work has been done on epidural analgesia, which is also a type of regional technique and attenuation of stress hormones is seen by the investigators with this form of analgesia. Epidural analgesia is an invasive procedure, which is expensive and requires expertise and equipment. It is not routinely practiced in our part of the world due to the above mentioned reasons. Epidural analgesia is used at AKUH, but it often less acceptable to patients as it is performed near the spinal cord and also because of the cost related issue.

Therefore the rational of this study is to observe, if a less expensive, easy to perform and safer form of regional analgesia like TAP block has an inhibitory effect on the surgical response or not. If favorable results are seen with TAP block, it can be incorporated in the practice guidelines of pain management for abdominal hysterectomies and related surgeries.

Primary Objective

This study is designed to test the hypothesis that the TAP block, as part of a multimodal analgesic regimen, would attenuate stress response after TAH when compared with placebo. An ultrasound (US)-guided TAP block will be performed before surgical incision.

Venous blood samples (20 ml) for metabolic and stress hormones, including cortisol and norepinephrine will be collected before anesthesia (T1) at the time of cannulation, and 30 minutes after incision(T2) 6hrs (T3)and 24 h (T4) after the surgery.

Secondary Objectives The investigators will observe any difference in postoperative pain by numeric rating score (NRS) and rescue analgesic demands by the reading on patient controlled analgesia pump, total opioid consumption and side effects like nausea, vomiting, sedation by scoring them.

Patient satisfaction score by scoring system

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective TAH via Pfannenstiel abdominal wall incision under general anaesthesia
* American Society of Anesthesiologists physical status I-II

Exclusion Criteria:

* Patients will be excluded if there is patient refusal to participate in the study, history of relevant drug allergy, or medical therapies considered to result in tolerance to opioids, hysterectomy performed for malignancy or inability to use patient control analgesia (PCA) devise

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06-17 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Serum Cortisol | 12 hours after surgery
  Serum cortisol measured in µg/dL
Serum Norepinephrine | 12 hours after surgery
  Serum norepinephrine levels in pg/ml

SECONDARY OUTCOMES:
Pain Score | 12 hours after surgery
  Pain will be measure by a Numeric Rating Score at rest and on movement. Numeric Rating Score will be from 1 to 10 where 1 is no pain and 10 is the most severe pain
Rescue analgesia | 12 hours after surgery
  Number of times rescue analgesia was required
Total amount of opioid consumption | 12 hours after surgery
  Total consumption in milligrams from Patient controlled intravenous analgesia machine
Side effects | 12 hours after surgery
  Nausea, Vomiting and sedation

OTHER OUTCOMES:
Patient satisfaction | 24 hours after surgery
  7-point Likert scale (1=strongly disagree, 7=strong¬ly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Samina Ismail, Principal Investigator — Aga Khan University

REFERENCES:
- [Background] Stanley G, Appadu B, Mead M, Rowbotham DJ. Dose requirements, efficacy and side effects of morphine and pethidine delivered by patient-controlled analgesia after gynaecological surgery. Br J Anaesth. 1996 Apr;76(4):484-6. doi: 10.1093/bja/76.4.484. PMID 8652316
- [Background] Woodhouse A, Mather LE. The effect of duration of dose delivery with patient-controlled analgesia on the incidence of nausea and vomiting after hysterectomy. Br J Clin Pharmacol. 1998 Jan;45(1):57-62. doi: 10.1046/j.1365-2125.1998.00635.x. PMID 9489595
- [Background] Ng A, Swami A, Smith G, Davidson AC, Emembolu J. The analgesic effects of intraperitoneal and incisional bupivacaine with epinephrine after total abdominal hysterectomy. Anesth Analg. 2002 Jul;95(1):158-62, table of contents. doi: 10.1097/00000539-200207000-00028. PMID 12088961
- [Background] Nishiyama T, Yamashita K, Yokoyama T. Stress hormone changes in general anesthesia of long duration: isoflurane-nitrous oxide vs sevoflurane-nitrous oxide anesthesia. J Clin Anesth. 2005 Dec;17(8):586-91. doi: 10.1016/j.jclinane.2005.03.009. PMID 16427527
- [Background] Chae BK, Lee HW, Sun K, Choi YH, Kim HM. The effect of combined epidural and light general anesthesia on stress hormones in open heart surgery patients. Surg Today. 1998;28(7):727-31. doi: 10.1007/BF02484619. PMID 9697266
- [Background] Li Y, Zhu S, Yan M. Combined general/epidural anesthesia (ropivacaine 0.375%) versus general anesthesia for upper abdominal surgery. Anesth Analg. 2008 May;106(5):1562-5, table of contents. doi: 10.1213/ane.0b013e31816d1976. PMID 18420877
- [Background] Yokoyama M, Itano Y, Katayama H, Morimatsu H, Takeda Y, Takahashi T, Nagano O, Morita K. The effects of continuous epidural anesthesia and analgesia on stress response and immune function in patients undergoing radical esophagectomy. Anesth Analg. 2005 Nov;101(5):1521-1527. doi: 10.1213/01.ANE.0000184287.15086.1E. PMID 16244024
- [Background] Ozyuvaci E, Altan A, Karadeniz T, Topsakal M, Besisik A, Yucel M. General anesthesia versus epidural and general anesthesia in radical cystectomy. Urol Int. 2005;74(1):62-7. doi: 10.1159/000082712. PMID 15711112
- [Background] Schricker T, Berroth A, Pfeiffer U, Schreiber M, Malik E, Schmidt M, Goertz A, Georgieff M. Influence of vaginal versus abdominal hysterectomy on perioperative glucose metabolism. Anesth Analg. 1996 Nov;83(5):991-5. doi: 10.1097/00000539-199611000-00016. PMID 8895274
- [Background] Minhas MR, Kamal R, Afshan G, Raheel H. Knowledge, attitude and practice of parturients regarding Epidural Analgesia for labour in a university hospital in Karachi. J Pak Med Assoc. 2005 Feb;55(2):63-6. PMID 15813631
- [Background] Abrahams MS, Aziz MF, Fu RF, Horn JL. Ultrasound guidance compared with electrical neurostimulation for peripheral nerve block: a systematic review and meta-analysis of randomized controlled trials. Br J Anaesth. 2009 Mar;102(3):408-17. doi: 10.1093/bja/aen384. Epub 2009 Jan 26. PMID 19174373
- [Background] Rafi AN. Abdominal field block: a new approach via the lumbar triangle. Anaesthesia. 2001 Oct;56(10):1024-6. doi: 10.1046/j.1365-2044.2001.02279-40.x. No abstract available. PMID 11576144
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] Netter FH Back and Spinal Cord. In: Netter FH, ed. Atlas of Human Anatomy Summit. New Jersey, USA: The Ciba-Geigy Corporation, 1989:145-55.
- [Background] McDonnell JG, Curley G, Carney J, Benton A, Costello J, Maharaj CH, Laffey JG. The analgesic efficacy of transversus abdominis plane block after cesarean delivery: a randomized controlled trial. Anesth Analg. 2008 Jan;106(1):186-91, table of contents. doi: 10.1213/01.ane.0000290294.64090.f3. PMID 18165577
- [Background] O'Donnell BD, McDonnell JG, McShane AJ. The transversus abdominis plane (TAP) block in open retropubic prostatectomy. Reg Anesth Pain Med. 2006 Jan-Feb;31(1):91. doi: 10.1016/j.rapm.2005.10.006. No abstract available. PMID 16418039
- [Background] Carney J, McDonnell JG, Ochana A, Bhinder R, Laffey JG. The transversus abdominis plane block provides effective postoperative analgesia in patients undergoing total abdominal hysterectomy. Anesth Analg. 2008 Dec;107(6):2056-60. doi: 10.1213/ane.0b013e3181871313. PMID 19020158
- [Background] Brennan F, Carr DB, Cousins M. Pain management: a fundamental human right. Anesth Analg. 2007 Jul;105(1):205-21. doi: 10.1213/01.ane.0000268145.52345.55. PMID 17578977
- [Background] Kehlet H, Holte K. Review of postoperative ileus. Am J Surg. 2001 Nov;182(5A Suppl):3S-10S. doi: 10.1016/s0002-9610(01)00781-4. PMID 11755891
- [Background] Perkins FM, Kehlet H. Chronic pain as an outcome of surgery. A review of predictive factors. Anesthesiology. 2000 Oct;93(4):1123-33. doi: 10.1097/00000542-200010000-00038. No abstract available. PMID 11020770
- [Background] Taylor R Jr, Pergolizzi JV, Raffa RB, Munzi E. Opioids: pharmacology, clinical uses and adverse effects. In: Tvildiani D, Gegechkori K, eds. Opioids: Pharmacology, Clinical Uses and Adverse Effects. Hauppauge, NY: Nova Science Publishers, Inc.; 2012:75-94
- [Background] Hodges SC, Mijumbi C, Okello M, McCormick BA, Walker IA, Wilson IH. Anaesthesia services in developing countries: defining the problems. Anaesthesia. 2007 Jan;62(1):4-11. doi: 10.1111/j.1365-2044.2006.04907.x. PMID 17156220
- [Background] De Lima L, Sweeney C, Palmer JL, Bruera E. Potent analgesics are more expensive for patients in developing countries: a comparative study. J Pain Palliat Care Pharmacother. 2004;18(1):59-70. PMID 15148009
- [Background] Engquist A, Brandt MR, Fernandes A, Kehlet H. The blocking effect of epidural analgesia on the adrenocortical and hyperglycemic responses to surgery. Acta Anaesthesiol Scand. 1977;21(4):330-5. doi: 10.1111/j.1399-6576.1977.tb01227.x. PMID 906788
- [Background] Hebbard P, Fujiwara Y, Shibata Y, Royse C. Ultrasound-guided transversus abdominis plane (TAP) block. Anaesth Intensive Care. 2007 Aug;35(4):616-7. No abstract available. PMID 18020088
- [Background] Webster K. The transversus abdominis plane (TAP) block: Abdominal plane regional anaesthesia. Update Anaesth. 2008; 24:25-30
- [Background] Myles PS, Wengritzky R. Simplified postoperative nausea and vomiting impact scale for audit and post-discharge review. Br J Anaesth. 2012 Mar;108(3):423-9. doi: 10.1093/bja/aer505. Epub 2012 Jan 29. PMID 22290456
- [Background] Jankovic Z, Ahmad N, Ravishankar N, Archer F. Transversus abdominis plane block: how safe is it? Anesth Analg. 2008 Nov;107(5):1758-9. doi: 10.1213/ane.0b013e3181853619. No abstract available. PMID 18931248
- [Background] Rosario DJ, Jacob S, Luntley J, Skinner PP, Raftery AT. Mechanism of femoral nerve palsy complicating percutaneous ilioinguinal field block. Br J Anaesth. 1997 Mar;78(3):314-6. doi: 10.1093/bja/78.3.314. PMID 9135313
- [Background] Walker G. Transversus abdominis plane block: a note of caution! Br J Anaesth. 2010 Feb;104(2):265. doi: 10.1093/bja/aep387. No abstract available. PMID 20086069
- [Derived] Ismail S, Ahmed A, Hoda MQ, Asghar S, Habib A, Aziz A. Mid-axillary transversus abdominis plane block and stress response after abdominal hysterectomy: A randomised controlled placebo trial. Eur J Anaesthesiol. 2021 Jul 1;38(7):768-776. doi: 10.1097/EJA.0000000000001413. PMID 33399377